CLINICAL TRIAL: NCT04364464
Title: Investigation of Pharmacokinetics, Safety, and Tolerability of BAY 63-2521 in Male and Female Subjects With Renal Impairment and in Age- and Weight- Matched Healthy Subjects Following a Single Oral Dose of 1 mg BAY 63-2521 in a Single-center, Non-randomized, Non-controlled, Non-blinded, Observational Study With Group Stratification
Brief Title: Study on the Safety of BAY 63-2521, How it is Tolerated and the Way the Body Absorbs, Distributes and Gets Rid of the Study Drug Given as a Single Oral Dose of 1 mg Tablet in Participants With Renal Impairment and Healthy Participants Matched for Age-, Gender-, and Weight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15000; 2009-017685-23 (EudraCT Number)
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Clinical Pharmacology
MeSH Terms: interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Riociguat, healthy participants (Experimental): Participants with creatinine clearance (CLCR) >80 mL/min received a single dose of 1 mg (2 x 0.5 mg IR tablet) of riociguat in the fasted state
  Interventions: Drug: Riociguat (Adempas, BAY 63-2521)
- Riociguat, mild renal impairment (Experimental): Participants with CLCR 50-80 mL/min received a single dose of 1 mg (2 x 0.5 mg IR tablet) of riociguat in the fasted state
  Interventions: Drug: Riociguat (Adempas, BAY 63-2521)
- Riociguat, moderate renal impairment (Experimental): Participants with CLCR 30-<50 mL/min received a single dose of 1 mg (2 x 0.5 mg IR tablet) of riociguat in the fasted state
  Interventions: Drug: Riociguat (Adempas, BAY 63-2521)
- Riociguat, severe renal impairment (Experimental): Participants with CLCR <30 mL/min received a single dose of 1 mg (2 x 0.5 mg IR tablet) of riociguat in the fasted state
  Interventions: Drug: Riociguat (Adempas, BAY 63-2521)

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY 63-2521) — 0.5 mg riociguat as an immediate-release (IR) tablet

SUMMARY:
BAY 63-2521 is intended to be used for a disease that affects the blood flow through the lungs. Renal impairment is a common condition in patients with this disease. The goal of the study is to learn more about the safety of BAY 63-2521, how it is tolerated and the way the body absorbs, distributes and gets rid of the study dug given as a single oral dose of 1 mg tablet in participants with renal impairment and healthy participants matched for age-, gender-, and weight

ELIGIBILITY:
Inclusion criteria for all subjects:

* Male and female white subjects with 18 to ≤79 years of age, BMI between 18 and 34 kg/m^2
* Women without childbearing potential or with childbearing potential but only if the pregnancy test is negative and are under highly effective contraception

Inclusion criteria for subjects with renal failure:

- Stable renal disease, ie. a serum creatinine value determined at least 3 - 6 months before the pre-study visit was not allowed to vary by more than 20% from the serum creatinine value determined at the pre-study visit

Inclusion criteria for healthy subjects:

- Mean age and body weight not allowed to vary by more than +/- 10 years and +/- 10 kg from the subjects with renal impairment, respectively

Exclusion criteria for all subjects:

* Febrile illness within 1 week before the start of the study
* Hypersensitivity to riociguat and / or to inactive constituents
* Smoking

Exclusion criteria for subjects with renal failure:

* Resting heart rate in the awake subject below 45 BPM or above 90 BPM
* Acute renal failure or nephritis
* Any organ transplant
* Diastolic blood pressure (DBP) >100 mmHg and / or systolic blood pressure (SBP) >180 mmHg
* Hemoglobin <8 g/dL, Proteinuria >8 g/24 hours, Serum albumin <30 g/L, Platelet count <100 x 109/L
* History of bleeding within the past 3 months
* Diabetes mellitus with a fasting blood glucose >220 mg/dL or HbA1c >10%
* Concomitant use of any medication except medications necessary for the treatment of the kidney disease or related complications
* Concomitant use of phosphodiesterase-5 inhibitors, endothelin receptor antagonists (ERAs, eg bosentan), intravenous or inhalative prostacyclins, or nitrates
* Concomitant use of potent CYP3A4 inhibitors

Exclusion criteria for healthy subjects:

* Conspicuous findings in medical history or pre-study examination
* History of relevant diseases of vital organs, central nervous system, or other organs
* SBP below 100 mmHg or above 145 mmHg and / or DBP above 95 mmHg
* Regular daily consumption of more than 1 liter of usual beer or the equivalent quantity of approximately 40 g of alcohol in another form

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02-19 (Actual); Primary Completion 2011-03-17 (Actual); Study Completion 2011-09-20 (Actual)

PRIMARY OUTCOMES:
AUC | Pre-dose up to 72 hours post-dose
  Area under the plasma concentration vs time curve from zero to infinity for total (bound and unbound) drug after single dose for BAY 63-2521 and its metabolite M1 (BAY 60-4552)
Cmax | Pre-dose up to 72 hours post-dose
  Maximum total (bound and unbound) drug concentration in plasma after single dose administration for BAY 63-2521 and its metabolite M1
t½ | Pre-dose up to 72 hours post-dose
  Half-life associated with the terminal slope for BAY 63-2521 and its metabolite M1
fu | From 2 hours post-dose up to 24 hours post-dose
  Fraction unbound for BAY 63-2521 and its metabolite M1
AUCu | From 2 hours post-dose up to 24 hours post-dose
  AUC for unbound drug for BAY 63-2521 and its metabolite M1
Cmax,u | From 2 hours post-dose up to 24 hours post-dose
  Cmax for unbound drug for BAY 63-2521 and its metabolite M1

SECONDARY OUTCOMES:
AUC/D | Pre-dose up to 72 hours post-dose
  AUC divided by dose for BAY 63-2521 and its metabolite M1
AUCnorm | Pre-dose up to 72 hours post-dose
  AUC divided by dose per kg body weight for BAY 63-2521 and its metabolite M1
AUCu,norm | From 2 hours post-dose up to 24 hours post-dose
  AUCnorm for unbound drug for BAY 63-2521 and its metabolite M1
AUC(0-tlast) | Pre-dose up to 72 hours post-dose
  AUC from time 0 to the last data point for BAY 63-2521 and its metabolite M1
Cmax/D | Pre-dose up to 72 hours post-dose
  Cmax divided by dose for BAY 63-2521 and its metabolite M1
Cmax,norm | Pre-dose up to 72 hours post-dose
  Cmax divided by dose per kg body weight for BAY 63-2521 and its metabolite M1
Cmax,u,norm | From 2 hours post-dose up to 24 hours post-dose
  Cmax,norm for unbound drug for BAY 63-2521 and its metabolite M1
tmax | Pre-dose up to 72 hours post-dose
  Time to reach Cmax (in case of two identical Cmax values, the first tmax was used) for BAY 63-2521 and its metabolite M1
MRT | Pre-dose up to 72 hours post-dose
  Mean residence time for BAY 63-2521 and its metabolite M1
CL/F | Pre-dose up to 72 hours post-dose
  Total body clearance of drug calculated after extravascular administration (eg apparent oral clearance) for BAY 63-2521 and its metabolite M1
CLu/F | From 2 hours post-dose up to 24 hours post-dose
  CL/F for unbound drug for BAY 63-2521 and its metabolite M1
Vz/F | Pre-dose up to 72 hours post-dose
  Apparent volume of distribution during terminal phase after extravascular administration for BAY 63-2521 and its metabolite M1
AE,ur | From 24 hours prior to drug administration up to 72 hours post-dose
  Amount of (total) drug excreted in urine for BAY 63-2521 and its metabolite M1
CLR | From 24 hours prior to drug administration up to 72 hours post-dose
  Renal body clearance of drug for BAY 63-2521 and its metabolite M1
Number of participants with adverse events | Approximately 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/